CLINICAL TRIAL: NCT05257642
Title: Testing the Usability of the REThink Game and the Efficacy of Its Main Game-based ER Strategies on the Stress Reactivity of Children and Adolescents
Brief Title: Testing the Efficacy of REThink Main Game-based ER Strategies on the Stress Reactivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Collaborators: The Executive Agency for Higher Education, Research, Development and Innovation Funding (Other)
Responsible Party: Principal Investigator, Oana David, Professor Ph.D, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: REThinkEMOTIONS
Record Dates: First submitted 2022-02-16; First posted 2022-02-25 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2022-11

CONDITIONS: Emotion Regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cognitive Change Groups (Experimental): The participants in this group will complete the pre-test measurements, then they will receive a level of the REThink Game that focuses on cognitive change. After playing the game they will receive an experimental task Cyberball and complete the post-test measurements.
  Interventions: Other: REThink Game
- Mindfulness Groups (Experimental): The participants in this group will complete the pre-test measurements, then they will receive a level of the REThink Game that focuses on mindfulness and relaxation. After playing the game they will receive an experimental task Cyberball and complete the post-test measurements
  Interventions: Other: REThink Game
- Positive bias Group (Experimental): The participants in this group will complete the pre-test measurements, then they will receive a level of the REThink Game that focuses on problem-solving. After playing the game they will receive an experimental task Cyberball and complete the post-test measurements
  Interventions: Other: REThink Game
- Control Group (No Intervention): The participants in this group will complete the pre-test measurements, then they will receive an experimental task Cyberball and complete the post-test measurements

INTERVENTIONS:
Other: REThink Game — REThink is a online therapeutic game developed by David and collaborators (2018), proved to be an efficient intervention to reduce emotional symptoms of children and adolescents.
  Arms: Cognitive Change Groups; Mindfulness Groups; Positive bias Group

SUMMARY:
This activity will aim to test the comparative efficacy of the main game-based emotion-regulation abilities training of the REThink online game: cognitive change, biofeedback and problem-solving in reducing stress reactivity of the children and adolescents

DETAILED DESCRIPTION:
Children included in this study (aged 8-16 years, G*Power estimated N=98) will be allocated to one of the three experimental conditions (cognitive change, biofeedback and problem-solving game based training based on the REThink online game levels), or no intervention Control condition. All children will be exposed afterwards to psychosocial stress in the form of peer rejection "ball toss" task. It will be measure both game-based skills outcomes, and EMA stress reactivity outcomes.

ELIGIBILITY:
Inclusion Criteria:

children and adolescents between 8 and 16 years provided written parental consent

Exclusion Criteria:

Intellectual disability or physical limitations precluded the use of the computer program

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 146 (Actual)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Levels of rational and irrational beliefs | Pre-intervention (one week before the intervention)
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Changes in rational and irrational beliefs | Post-intervention (one week afterthe intervention)
  The Child and Adolescent Scale of Irrationality (CASI, Bernard & Cronan, 1999) will be used in order to test irrational/rational beliefs as a mechanism of change. Children and adolescents were asked to express their agreement/disagreement with the 28 statements on a 5-point Likert-type scale, from 1 ("strong disagreement") to 5 ("strong agreement")
Levels of mindfulness | Pre-intervention (one week before the intervention)
  The Mindfulness Awarness Attention Scale - Child version (MAAS-C, Lawlor, Reichl & Zumbo, 2014) is a 15-items questionnaire rated on a 6 points Likert scale from "almost never" to "almost every time" where higher scores means higher mindfulness.
Changes in levels of mindfulness | Post-intervention (one week afterthe intervention)
  The Mindfulness Awarness Attention Scale - Child version (MAAS-C, Lawlor, Reichl & Zumbo, 2014) is a 15-items questionnaire rated on a 6 points Likert scale from "almost never" to "almost every time" where higher scores means higher mindfulness.
Levels of well-being | Pre-intervention (one week before the intervention)
  WHO-5 Well-being Index
Changes in levels of well-being | Post-intervention (one week afterthe intervention)
  WHO-5 Well-being Index
Levels of emotion-regulation | Pre-intervention (one week before the intervention)
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Changes in levels of emotion-regulation | Post-intervention (one week afterthe intervention)
  The Emotion Regulation Index for Children and Adolescents (ERICA; Biesecker & Easterbrooks, 2001). It is a 13-item on a five-point Likert scale, from 0 "strong disagreement" to 5"strong agreement" where higher scores represent better emotional regulation abilities,
Level of distress | Pre-intervention (one week before the intervention)
  Measured with Profile of Emotional Distress
Changes in level of distress | Post-intervention (one week afterthe intervention)
  Measured with Profile of Emotional Distress
Children Emotional Abilities | Pre-intervention (one week before the intervention)
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.
Changes in children Emotional Abilities | Post-intervention (one week afterthe intervention)
  The Cognitive Emotion Regulation Questionnaire - Short (Garnefski & Kraaij, 2006) is an 18-item self-report scale that measures a total of nine different cognitive coping strategies, each addressed by two items.

CONTACTS AND LOCATIONS:
Overall Officials: Oana David, Ph.D, Principal Investigator — Babes-Bolyai University
Locations (1):
- Babes-Bolyai University, Cluj-Napoca, Romania

IPD SHARING:
Plan to Share IPD: No